CLINICAL TRIAL: NCT01004211
Title: A Phase III Prospective Multicenter Randomized Comparison of Transurethral Resection by Mean of White Light and Narrow Band Imaging.
Brief Title: Prospective Randomized Comparison of Transurethral Resection by Mean of White Light and Narrow Band Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paolo Puppo (Other)
Responsible Party: Sponsor-Investigator, Paolo Puppo, MD, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Organization: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IST-NBI-2009
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Non Muscle Invasive Bladder Cancer
Keywords: bladder cancer; recurrence
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard transurethral resection (Active Comparator): Patients will be submitted to standard white light transurethral resection and/or cold cup biopsies of all visible lesions known or suspected to be bladder cancer; 6 random cold cup biopsies from healthy mucosa of bladder trigone, anterior, posterior and lateral walls will be taken in case of a second transurethral resection of newly diagnosed high grade non muscle invasive bladder cancer or of recurrent high grade non muscle invasive bladder cancer
  Interventions: Procedure: Standard transurethral resection
- Narrow band imaging transurethral resection (Experimental): The system will be switched to narrow band imaging by simply pushing a button. Transurethral resection and/or cold cup biopsies of all visible lesions known or suspected to be bladder cancer will be performed; 6 random cold cup biopsies from healthy mucosa of bladder trigone, anterior, posterior and lateral walls will be taken in case of a second transurethral resection of newly diagnosed high grade non muscle invasive bladder cancer or of recurrent high grade non muscle invasive bladder cancer.
  Interventions: Procedure: Narrow band imaging transurethral resection

INTERVENTIONS:
Procedure: Narrow band imaging transurethral resection — Transurethral resection of bladder lesion by mean of narrow band imaging
  Arms: Narrow band imaging transurethral resection
Procedure: Standard transurethral resection — Transurethral resection of bladder lesion by mean of standard white light
  Arms: Standard transurethral resection

SUMMARY:
To date, fluorescence and narrow band imaging cystoscopy have been tested in many prospective within patient trials but only as an "add on" procedure. This results in a bias that does not allow to determine the real impact of such innovative technologies on bladder cancer management. Hereby we propose the first prospective randomized trial which compares narrow band imaging trans urethral resection as a stand alone procedure versus white light transurethral resection. The primary end point is to assess the recurrence rate of bladder cancer lesions with each treatment modality. The study is designed to disclose an inferior recurrence rate (estimated 10%) in the group treated by narrow band imaging transurethral resection respect to the control group, treated by standard transurethral resection.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be older than 18 years of age and female patients who are pregnant, breast feeding or not on adequate contraceptive measures will be excluded.
* All patients will provide a written informed consent prior to the study.
* Consecutive patients from 2 centers in Liguria (National Institute for Cancer Research - Genova and Centro Urologico di Eccellenza ASL 1 - Imperia) with overt or suspected non muscle invasive bladder cancer, including Cis detected by mean of random biopsies or a positive urinary cytology, will be included in the study and randomized to 2 treatments A, B arms.

Exclusion Criteria:

* Patients with muscle invasive bladder cancer will be excluded.
* Patients submitted to immediate radical cystectomy after transurethral resection, irrespective of the clinical stage, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2009-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Recurrence free survival rate | One year

SECONDARY OUTCOMES:
Detection rate | At the end of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Puppo, MD, Principal Investigator — National Institute for Cancer Research, Genoa, Italy
Locations (2):
- Italy (2):
  - National Institute for Cancer Research (IST), Genoa
  - Centro Urologico di Eccellenza ASL 1, Imperia

REFERENCES:
- [Background] Naselli A, Introini C, Bertolotto F, Spina B, Puppo P. Narrow band imaging for detecting residual/recurrent cancerous tissue during second transurethral resection of newly diagnosed non-muscle-invasive high-grade bladder cancer. BJU Int. 2010 Jan;105(2):208-11. doi: 10.1111/j.1464-410X.2009.08701.x. Epub 2009 Jun 22. PMID 19549255
- [Result] Naselli A, Introini C, Bertolotto F, Spina B, Puppo P. Feasibility of transurethral resection of bladder lesion performed entirely by means of narrow-band imaging. J Endourol. 2010 Jul;24(7):1131-4. doi: 10.1089/end.2010.0042. PMID 20509796
- [Result] Naselli A, Introini C, Timossi L, Spina B, Fontana V, Pezzi R, Germinale F, Bertolotto F, Puppo P. A randomized prospective trial to assess the impact of transurethral resection in narrow band imaging modality on non-muscle-invasive bladder cancer recurrence. Eur Urol. 2012 May;61(5):908-13. doi: 10.1016/j.eururo.2012.01.018. Epub 2012 Jan 20. PMID 22280855